CLINICAL TRIAL: NCT05272501
Title: CAlming Touch for People With Agitation or Other Behavioural Symptoms of DEMentia - A Randomized Feasibility Trial
Acronym: CADEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Copenhagen (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 200576
Record Dates: First submitted 2021-12-17; First posted 2022-03-09 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Dementia; Agitation,Psychomotor
MeSH Terms: conditions — Dementia; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calming Touch (Experimental): The calming treatment consists of deep pressure massage and gentle facilitation. The therapist works with the vertical axis, center, respiration, body boundaries and the feet.
  Interventions: Behavioral: Calming Touch
- Usual care (No Intervention): The usual care group may participate in usual activities at the nursing home e.g. physio- and occupational therapy, listening to calming music, holdning hands with care-takers.

INTERVENTIONS:
Behavioral: Calming Touch — The calming treatment consists of deep pressure massage and gentle facilitation. The therapist works with the vertical axis, center, respiration, body boundaries and the feet.
  Arms: Calming Touch

SUMMARY:
Dementia is an increasing health challenge among elderly citizens in Denmark. An estimated 87,000 Danes live with dementia, and this number is expected to increase to 130,000 in 2030. Psychiatric symptoms and behavioral changes decrease quality of life for patients and their spouses and is a challenge for caretakers. Behavior changes include agitation which can be divided in four sub-groups: 1) physical aggression, 2) physical non-aggression, 3) verbal aggression, and 4) verbal non-aggression. Pharmaceutical management of behavioral changes is common and may be associated with negative side-effects including drowsiness and falls. Though non-pharmaceutical interventions such as music, massage and social activities have been recommended the underlying evidence is limited. In this randomized feasibility trial, we will investigate the feasibility and acceptability of therapeutic touch aiming to reduce agitated behavior in people living with dementia in a nursing home that specializes in the care of people living with severe dementia.

The success criteria of this randomized feasibility trial are as follows:

1. Nursing home residents can be recruited and accept the treatment 'CAlming Touch for People with Agitation or Other Behavioral Symptoms of DEMentia' (CADEM) and complete the feasibility project's test protocol.
2. The treatment concept, which involves the nursing staff in charge of the follow-up treatment, can be implemented in practice.
3. The treatment (CADEM) shows a tendency towards less restless and aggressive behavior for demented citizens evaluated based on a validated measuring tool.

ELIGIBILITY:
Inclusion Criteria:

* Citizens who are residents of the care center due to dementia
* Citizens living at a care center in Naestved Municipality
* Demented citizens who exhibit agitated / aggressive behavior (nursing staff observe whether the citizen exhibits agitated behavior within at least one of the subgroups

Exclusion Criteria:

* Citizens in palliative care
* Citizens who have received BBAUM treatment within the last month

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Change in Cohen-Mansfield Agitation Inventory (CMAI) from baseline to 4, 8, and 12 weeks after baseline. | CMAI will be performed 2 weeks before baseline, at baseline, and 4, 8, and 12 weeks post baseline.
  The Cohen-Mansfield Agitation Inventory (CMAI; Cohen-Mansfield, 1986) is a 29-item questionnaire designed to measure the types and frequencies of agitated behaviors exhibited by elderly nursing home residents

SECONDARY OUTCOMES:
The Erlangen Test for Activities of Daily Living (E-ADL-Test) | The E-ADL-Test will be performed at baseline, and 4, 8, and 12 weeks post baseline.
  The Erlangen Test of Activities of Daily Living (E-ADL-Test) consists of five items: pouring a drink, cutting a piece of bread, opening a small cupboard, washing hands and tying a bow. Each test item underwent standardized evaluation on a scale of 0 to 6.
Hair cortisol levels | Hair samples will be collected at baseline, and 4, 8, and 12 weeks post baseline.
  Hair samples will be collected and cortisol levels will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Jonna Jensen, Ass. Prof., Principal Investigator — University College Copenhagen
Locations (1):
- Distrikt Oest., Næstved, Denmark

IPD SHARING:
Plan to Share IPD: No